CLINICAL TRIAL: NCT01127737
Title: Warning Signs of Squamous Cell Carcinoma and Prevention of SCC by at Risk Organ Transplant Recipients
Acronym: SCCs in OTRs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: JKR-090607
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Squamous Cell Carcinoma
Keywords: SCCs; Squamous Cell Carcinoma; Skin Self Exam; SSE; Organ Transplant; Performance of SSE with our written educational intervention; Time after organ transplantation to deliver intervention; Evaluate internation information
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Behavioral: Placebo
- Intervention (Active Comparator): Educational intervention consisting of a mnemonic and a workbook used by kidney transplant recipients (KTRs) to assist with early detection of SCCs.
  Interventions: Behavioral: Educational Intervention; Behavioral: Placebo

INTERVENTIONS:
Behavioral: Educational Intervention — Mnemonic and a workbook used by kidney transplant recipients to assist with early early detection of SCCs.
  Arms: Intervention
Behavioral: Placebo — Completed surveys

SUMMARY:
Using focus group and cognitive interviews with organ transplant recipients, the investigators developed interactive workbooks: a) prevention by sun protection b) early detection by skin self-examination (SSE). The investigators hypothesis is if the patient learns by acquiring skills in a favorable environment, then the patient may reduce their anxiety, enhance self-efficacy and perform self-management by SSE and sun protection. The investigators also evaluate existing internet sources of primary and secondary prevention of skin cancer for organ transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* People with a history of solid organ transplantation within the last 2 years
* Speaks English
* Can see to do SSE, capable of seeing to read a newspaper
* Stable health, patients report a general state of well being

Exclusion Criteria:

* Unable to speak English
* Insufficient vision to see their own skin as determined by their ability to read a newspaper
* Comorbid debilitating disease
* Dementia or insufficient cognitive skills to follow instructions provided at a sixth grade language level.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P West, PhD, Study Chair — Northwestern University; June K Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Robinson JK, Turrisi R, Mallett KA, Stapleton J, Boone SL, Kim N, Riyat NV, Gordon EJ. Efficacy of an educational intervention with kidney transplant recipients to promote skin self-examination for squamous cell carcinoma detection. Arch Dermatol. 2011 Jun;147(6):689-95. doi: 10.1001/archdermatol.2011.10. Epub 2011 Feb 21. PMID 21339418
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Northwestern University's kidney transplant recipient population. Participants were returning for routine care to their nephrologists 1 to 1.2 years or 3 to 7 years after transplantation.
Groups:
- Control: Control group received only intiial assessment at the time of physician visit and education as usually provided during the physician visit.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 37 | 38
Completed | 37 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Median (Full Range); unit: years] | 58 [25 to 74] | 61 [32 to 76] | 60 [25 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Control and Intervention Participants on Skin Self-examination Performance at Follow-up 1 Month After Intervention
Description: The number of control and intervention participants who checked their skin for cancer within the 1 month after the study visit.
Time Frame: 1 month
Population: Per protocol
Measure: Number; unit: Participants
Groups:
- Intervention: Educational intervention consisting of a mnemonic and a workboook
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 38 | 37
Participants | 34 | 8

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

LIMITATIONS AND CAVEATS:
* Small sample at a single center for a limited period of follow-up
* The dermatologists' assessment of the participants' concerning lesions was not performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No